CLINICAL TRIAL: NCT00262795
Title: Fludarabine Versus Chlorambucil in First Line Therapy of Elderly Patients (More Than 65 Years) With Advanced Chronic Lymphocytic Leukemia
Brief Title: Fludarabine or Chlorambucil as First-Line Therapy in Treating Older Patients With Previously Untreated Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLL5; EU-20557; MEDAC-GCLLSG-CLL5; GCLLSG-73
Record Dates: First submitted 2005-12-06; First posted 2005-12-07 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — fludarabine; Chlorambucil

ARMS (2):
- F (Experimental): Fludarabine
  Interventions: Drug: Fludarabine
- CLB (Active Comparator): Chlorambucil
  Interventions: Drug: Chlorambucil

INTERVENTIONS:
Drug: Fludarabine — Fludarabine i.v. (25 mg/m2/d, d1-5) q28d; max 6 cycles
  Arms: F
Drug: Chlorambucil — Chlorambucil p.o. (0,4 mg - max. 0,8 mg/kg/d, d1) q15d, max. 12 month
  Arms: CLB

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and chlorambucil, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not yet known whether fludarabine is more effective than chlorambucil in treating chronic lymphocytic leukemia.

PURPOSE: This randomized phase III trial is studying fludarabine to see how well it works as first-line therapy compared to chlorambucil in treating older patients with previously untreated chronic lymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the overall and progression-free survival of older patients with previously untreated chronic lymphocytic leukemia treated with fludarabine vs chlorambucil.
* Compare the duration of remission in patients treated with these regimens.

Secondary

* Compare the incidence of toxicity, especially infections, in patients treated with these regimens.
* Compare the quality of life in patients treated with these regimens.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive fludarabine IV on days 1-5. Treatment repeats every 28 days for up to 6 courses.
* Arm II: Patients receive oral chlorambucil on day 1. Treatment repeats every 15 days for up to 12 months.

PROJECTED ACCRUAL: A total of 205 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Confirmed diagnosis of chronic lymphocytic leukemia, meeting any of the following staging criteria:

  * Binet stage A with B symptoms
  * Binet stage B or C, meeting 1 of the following criteria:

    * Rapid disease progression
    * Enlarged lymph nodes and organs
    * Severe B symptoms
* Previously untreated disease

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* No thrombocytopenia
* No autoimmune hemolytic anemia

Hepatic

* Not specified

Renal

* Not specified

Other

* No severe organ dysfunction
* No other prior or concurrent neoplasm

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Ages: 65 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 206 (Actual)
Dates: Start 2003-09; Primary Completion 2005-01 (Actual); Study Completion 2005-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hallek, MD, Study Chair — Medizinische Universitaetsklinik I at the University of Cologne
Locations (88):
- Hanuschkrankenhaus, Vienna, Austria
- Germany (87):
  - Klinikum St. Marien, Amberg
  - Gemeinschaftspraxis Fuer Innere Medizin, Haematologie Und Internistische Onkologie, Ansbach
  - Zentralklinikum Augsburg, Augsburg
  - Humaine - Clinic, Bad Saarow
  - Krankenhaus Hohe Warte Mediziniche Klinik, Bayreuth
  - Onkologisches Versorgungszentrum Friedrichshain, Berlin
  - Internistische Gemeinschaftspraxis - Berlin, Berlin
  - Charite - Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Charite - Campus Virchow Klinikum, Berlin
  - Saint Josef - Hospital Bochum, Bochum
  - Praxis Dres. F.& G. Doering, Bremen
  - Medizinische Universitaetsklinik I at the University of Cologne, Cologne
  - Onkologische Schwerpunktpraxis, Cottbus
  - Onkologische Gemeinschaftspraxis - Dresden, Dresden
  - Krankenhaus Benrath, Düsseldorf
  - Hans - Susemihl - Krankenhaus, Emden
  - Kreiskrankenhaus Erding, Erding
  - Internistische/Onkologische Praxis - Erfurt, Erfurt
  - Helios Klinikum Erfurt, Erfurt
  - Onkologische Schwerpunkt Praxis, Erlangen
  - Universitaetsklinikum Essen, Essen
  - Evangelisches Krankenhaus Essen Werden, Essen
  - Gemeinschaftspraxis - Freiburg, Freiburg im Breisgau
  - Klinikum Garmisch - Partenkirchen, Garmisch-Partenkirchen
  - Gemeinschaftspraxis Innere Medizin Hämatologie/Onkologie - Gera, Gera
  - Internistische Praxis - Gerlingen, Gerlingen
  - Internistische Praxisgemeinschaft, Germering
  - Universitaetsklinikum Goettingen, Göttingen
  - Internistisch-Haematologische Gemeinschaftspraxis - Gustrow, Güstrow
  - Internistische Praxis - Halle, Halle
  - Internistische Gemeinschaftspraxis - Halle, Halle
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - St. Marien-Hospital Hamm - Klinik Knappenstrasse, Hamm
  - Schwerpunktpraxis Haematologie/Onkologie - Hannover, Hanover
  - Eichsfeld Klinikum gGmbH, Heiligenstadt
  - Medizinischen Klinik Dr. R. Schindlbeck, Herrsching am Ammersee
  - Oncological Specialist Practice, Hildesheim
  - Universitaetsklinikum des Saarlandes, Homburg
  - Clinic for Bone Marrow Transplantation and Hematology and Oncology, Idar-Oberstein
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Staedt Klinikum Karlsruhe GGMBH, Karlsruhe
  - Internistische Gemeinschaftspraxis - Kassel, Kassel
  - Staedtische Krankenhaus Kiel, Kiel
  - Krankenhaus Maria-Hilf Krefeld, Krefeld
  - Internistische Onkologische Praxis - Kronach, Kronach
  - Internistische Praxis - Landshut, Landshut
  - Klinikum Lippe - Lemgo, Lemgo
  - Internistische Praxis - Ludwigsburg, Ludwigsburg
  - Kreiskrankenhaus Luedenscheid, Lüdenscheid
  - III Medizinische Klinik Mannheim, Mannheim
  - Regional Hospital Munchberg, Munchber
  - Klinikum Innenstadt, Munich
  - Krankenhaus Muenchen Schwabing, Munich
  - Hamatologische Schwerpunktpraxis, Munich
  - Munich Oncologic Practice at Elisenhof, Munich
  - Klinikum der Universitaet Muenchen - Grosshadern Campus, Munich
  - Staedtisches Krankenhaus Muenchen - Harlaching, Munich
  - Klinikum Rechts Der Isar - Technische Universitaet Muenchen, Munich
  - Hamatologie/Onkologie Praxisgemeinschaft - Munchen, München
  - Haematologisch-onkologische Gemeinschaftspraxis - Muenster, Münster
  - Onkologische Schwerpunktpraxis Dr. Schmidt, Neunkirchen
  - Praxis fuer Haematologie und Interne Onkologie, Norderstedt
  - Praxisklinik fuer Innere Medizin - Nuernberg, Nuremberg
  - Klinikum Nuernberg - Klinikum Nord, Nuremberg
  - Internistische Gemeinschaftspraxis - Oberstaufen, Oberstaufen
  - Internistische Gemeinschaftspraxis - Offenbach, Offenbach
  - Internistische Gemeinschaftspraxis - Oldenburg, Oldenburg
  - Klinikum Ernst Von Bergmann, Postdam
  - Haematologische/Onkologische Schwerpunktpraxis - Rostock, Rostock
  - Klinik und Poliklinik fuer Innere Medizin - Universitaet Rostock, Rostock
  - Internistische Schwerpunktpraxis, Rüsselsheim am Main
  - Schwerpunktpraxis Fuer Haematologie Und Onkologie, Saarbruecke
  - Internistische Gemeinschaftspraxis - Saarbruecken, Saarbrücken
  - Caritasklinik St. Theresia, Saarbrücken
  - Kliniken Landkreis Sigmaringen GMBH, Sigmaringen
  - Internistische Gemeinschaftspraxis - Stuttgart, Stuttgart
  - Marienhospital Stuttgart, Stuttgart
  - Haematologische Praxis, Stuttgart
  - Klinik fuer Onkologie - Katharinenhospital Stuttgart, Stuttgart
  - Onkologische Gemeinschaftspraxis - Trier, Trier
  - Krankenanstalt Mutterhaus der Borromaerinnen, Trier
  - Southwest German Cancer Center at Eberhard-Karls-University, Tübingen
  - Universitaetsklinikum Ulm, Ulm
  - St. Marien Hospital, Vechta
  - Gemeinschaftspraxis, Worms
  - Kliniken St. Antonius, Wuppertal
  - Hamatologisch - Onkologische Praxis Wurzburg, Würzburg

REFERENCES:
- [Background] Eichhorst BF, Fischer K, Fink AM, Elter T, Wendtner CM, Goede V, Bergmann M, Stilgenbauer S, Hopfinger G, Ritgen M, Bahlo J, Busch R, Hallek M; German CLL Study Group (GCLLSG). Limited clinical relevance of imaging techniques in the follow-up of patients with advanced chronic lymphocytic leukemia: results of a meta-analysis. Blood. 2011 Feb 10;117(6):1817-21. doi: 10.1182/blood-2010-04-282228. Epub 2010 Dec 7. PMID 21139079
- [Background] Cramer P, Bahlo J, Eichhorst B, Fischer K, Hallek M. Extramedullary manifestations of chronic lymphocytic leukaemia are not unusual. Leuk Res. 2014 Mar;38(3):284-5. doi: 10.1016/j.leukres.2013.11.015. Epub 2013 Dec 1. No abstract available. PMID 24412156
- [Background] Goede V, Cramer P, Busch R, Bergmann M, Stauch M, Hopfinger G, Stilgenbauer S, Dohner H, Westermann A, Wendtner CM, Eichhorst B, Hallek M; German CLL Study Group. Interactions between comorbidity and treatment of chronic lymphocytic leukemia: results of German Chronic Lymphocytic Leukemia Study Group trials. Haematologica. 2014 Jun;99(6):1095-100. doi: 10.3324/haematol.2013.096792. Epub 2014 Feb 28. PMID 24584349
- [Background] Sachanas S, Pangalis GA, Fink AM, Bahlo J, Fischer K, Levidou G, Kyrtsonis MC, Bartzi V, Vassilakopoulos TP, Kalpadakis C, Koulieris E, Moschogiannis M, Yiakoumis X, Tsirkinidis P, Angelopoulou MK, Eichhorst B, Hallek M. Small Lymphocytic Lymphoma: Analysis of Two Cohorts Including Patients in Clinical Trials of the German Chronic Lymphocytic Leukemia Study Group (GCLLSG) or in "Real-Life" Outside of Clinical Trials. Anticancer Res. 2019 May;39(5):2591-2598. doi: 10.21873/anticanres.13382. PMID 31092457
- [Result] Eichhorst BF, Busch R, Stilgenbauer S, Stauch M, Bergmann MA, Ritgen M, Kranzhofer N, Rohrberg R, Soling U, Burkhard O, Westermann A, Goede V, Schweighofer CD, Fischer K, Fink AM, Wendtner CM, Brittinger G, Dohner H, Emmerich B, Hallek M; German CLL Study Group (GCLLSG). First-line therapy with fludarabine compared with chlorambucil does not result in a major benefit for elderly patients with advanced chronic lymphocytic leukemia. Blood. 2009 Oct 15;114(16):3382-91. doi: 10.1182/blood-2009-02-206185. Epub 2009 Jul 15. PMID 19605849